CLINICAL TRIAL: NCT00404248
Title: Phase I/II Study of Intravenous Infusion of Tetra-o-Methyl Nordihydroguaiaretic Acid (EM-1421) in Subjects With Recurrent High Grade Glioma
Brief Title: Tetra-O-Methyl Nordihydroguaiaretic Acid in Treating Patients With Recurrent High-Grade Glioma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NABTT-0503 CDR0000515952; U01CA062475 (NIH); NABTT-0503
Record Dates: First submitted 2006-11-27; First posted 2006-11-28 (Estimated); Results first posted 2015-08-11 (Estimated); Last update posted 2019-03-06 (Actual); Status verified 2019-03

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: adult anaplastic astrocytoma; adult anaplastic oligodendroglioma; adult giant cell glioblastoma; recurrent adult brain tumor; adult glioblastoma; adult gliosarcoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Astrocytoma; Oligodendroglioma; Glioblastoma; Brain Neoplasms; Gliosarcoma | interventions — terameprocol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- With Enzyme-inducing antiseizure drugs (+EIASD) (Active Comparator): subjects on the +EIASD treatment arm were taking one of these antiseizure drugs: phenytoin, carbamazepine, phenobarbital, primidone and oxcarbazepine.
  Subjects will take terameprocol for 5 consecutive days each month by IV. Starting dose is 750mg/day. Dose escalation is 750, 1100, 1700, 2200, 3000, 4000, 5300, 7000, and 9300. NO intrasubject dose escalation.
  PK (pharmacological study) data will be collected on day one of cycle one infusion
  Interventions: Drug: terameprocol; Other: pharmacological study
- With Non enzyme-inducing antiseizure drugs (-EIASD) (Active Comparator): Subjects in the -EIASD group were either not being treated with antiseizure drugs or were taking ones that did not significantly induce hepatic enzymes such as gabapentin, lamotrigine, valproic acid, levetiracetam, tiagabine, topiramate, zonisamide and felbamate.
  Subjects will take terameprocol for 5 consecutive days each month by IV. Starting dose is 750mg/day. Dose escalation is 750, 1100, 1700, 2200, 3000, 4000, 5300, 7000, and 9300. NO intrasubject dose escalation.
  PK (pharmacological study) data will be collected on day one of cycle one infusion
  Interventions: Drug: terameprocol; Other: pharmacological study

INTERVENTIONS:
Drug: terameprocol — terameprocol will be given IV 5 consecutive days every 28 days. Starting dose 750mg/day. Cohorts of 3pts. A Dose Limiting Toxicity (DLT) target rate of Less than or equal to 33%. Dose levels: 750, 1100, 1700, 2200, 3000, 4000, 5300, 7000, 9300 mg.
  Other Names: EM-1421
Other: pharmacological study — All pts on both arms will have pks, blood collections. 5ml of blood will be drawn on Cycle 1 day 1, Cycle 1 Day 5, Cycle 2 day 1 and Cycle 2 day 5. A total of 10 samples will be drawn at each of these time points. 1hr pre-infusion, 15 min, 1hr, 1.15, 1.5, 2, 3,4,6 and 24hr post infusion.
  Other Names: PK

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as tetra-O-methyl nordihydroguaiaretic acid (EM-1421), work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing.

PURPOSE: This phase I/II trial is studying the side effects and best dose of EM-1421 and to see how well it works in treating patients with recurrent high-grade glioma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the maximum tolerated dose (MTD) of tetra-O-methyl nordihydroguaiaretic acid (EM-1421) in patients with recurrent high-grade glioma. (Phase I)
* Determine the response rate in patients treated with EM-1421 administered at the MTD. (Phase II)

Secondary

* Describe the pharmacokinetics of EM-1421 in these patients. (Phase I)
* Determine the effects of hepatic enzyme-inducing anticonvulsants on the pharmacokinetic profile of EM-1421 in these patients. (Phase I)
* Determine the toxicity of this drug in these patients. (Phase I)
* Assess the tolerability of this drug in these patients. (Phase I)
* Assess the antitumor activity of this drug, in terms of overall survival. (Phase I)
* Assess the overall survival of these patients. (Phase II)
* Assess the safety and tolerability of EM-1421 given at the MTD in these patients. (Phase II)

OUTLINE: This is a multicenter, phase I, dose-escalation study followed by a phase II, open-label study. Patients are stratified according to the use of cytochrome P450-inducing anticonvulsants (use of anticonvulsant drugs that induce hepatic metabolic enzymes vs use of anticonvulsant drugs that cause modest or no induction of hepatic metabolic enzymes or no use of anticonvulsant drugs).

* Phase I: Patients receive tetra-O-methyl nordihydroguaiaretic acid (EM-1421) IV on days 1-5. Treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of EM-1421 until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 3 of 6 patients experience dose-limiting toxicity.

* Phase II: Patients receive EM-1421 as in phase I at the MTD. Blood is collected on days 1 and 5 of courses 1 and 2 of treatment for pharmacokinetic studies.

After completion of study therapy, patients are followed every 2 months.

PROJECTED ACCRUAL: A total of 50 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed malignant glioma, including any of the following subtypes:

  * Anaplastic astrocytoma
  * Anaplastic oligodendroglioma
  * Glioblastoma multiforme
* Progressive or recurrent disease after radiation therapy with or without chemotherapy

  * Patients with a previous low-grade glioma that has progressed to biopsy-confirmed high-grade glioma after radiation therapy with or without chemotherapy are eligible
* Contrast-enhancing measurable disease by MRI or CT scan

PATIENT CHARACTERISTICS:

* Karnofsky performance status 60-100%
* Absolute neutrophil count ≥ 1,500/mm³
* Hemoglobin ≥ 9 g/dL
* Platelet count ≥ 100,000/mm³
* Creatinine ≤ 1.5 mg/dL
* Bilirubin ≤ 1.5 mg/dL
* Transaminases ≤ 4 times upper limit of normal
* Prothrombin Time (PT)/partial thromboplastin time (PTT) /international normalized ratio (INR) normal
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective barrier contraception during and for 2 months after completion of study treatment
* Mini Mental State Exam score ≥ 15
* No serious concurrent infection or medical illness that would impair the ability to safely receive study treatment
* No other prior or concurrent malignancy within the past 5 years except for curatively treated carcinoma in situ or basal cell carcinoma of the skin
* No known sensitivity to any of the study medication components (i.e., polyethylene glycol [PEG 300] and 2-hydroxypropyl β-cyclodextrin)

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* Recovered from prior therapy
* At least 3 months since prior radiation therapy
* At least 3 weeks since prior chemotherapy (6 weeks for nitrosoureas)
* At least 2 weeks since prior Federal Drug Administration (FDA)-approved noncytotoxic therapy (e.g., celecoxib or thalidomide)
* At least 3 weeks since prior investigational noncytotoxic agents
* At least 10 days since prior anticonvulsant drugs that induce hepatic metabolic enzymes, including any of the following:

  * Phenytoin
  * Carbamazepine
  * Phenobarbital
  * Primidone
  * Oxcarbazepine
  * Ethosuximide
* No other concurrent therapy for this tumor, including systemic chemotherapy or radiation therapy

  * Concurrent steroids allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2007-01; Primary Completion 2009-06 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stuart A. Grossman, MD, Study Chair — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (9):
- United States (9):
  - UAB Comprehensive Cancer Center, Birmingham, Alabama
  - H. Lee Moffitt Cancer Center and Research Institute at University of South Florida, Tampa, Florida
  - Winship Cancer Institute of Emory University, Atlanta, Georgia
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Josephine Ford Cancer Center at Henry Ford Hospital, Detroit, Michigan
  - Wake Forest University Comprehensive Cancer Center, Winston-Salem, North Carolina
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania

REFERENCES:
- [Result] Grossman SA, Ye X, Peereboom D, Rosenfeld MR, Mikkelsen T, Supko JG, Desideri S; Adult Brain Tumor Consortium. Phase I study of terameprocol in patients with recurrent high-grade glioma. Neuro Oncol. 2012 Apr;14(4):511-7. doi: 10.1093/neuonc/nor230. Epub 2012 Feb 8. PMID 22323663
- See also: Clinical trial summary from the National Cancer Institute's PDQ® database — https://clinicaltrials.gov/ct2/show/NCT00404248?term=NABTT+0503&rank=1

RESULTS

PARTICIPANT FLOW:
Recruitment Details: subjects were accrued 2007-2008 in outpatient clinic
Groups:
- Arm 1 Enzyme Inducing Antiseizure Drug (+ EIASD) Level 1: subjects on the +EIASD (Level 1) treatment arm were taking one of these antiseizure drugs: phenytoin, carbamazepine, phenobarbital, primidone and oxcarbazepine.
  Subjects will take terameprocol for 5 consecutive days each month by IV. Dose level 1= 750mg/day. NO intrasubject dose escalation.
  Pharmacokinetics (PK) data will be collected on day one of cycle one infusion
- Arm 2 +EIASD Level 2: subjects on the +EIASD (Level 2) treatment arm were taking one of these antiseizure drugs: phenytoin, carbamazepine, phenobarbital, primidone and oxcarbazepine.
  Subjects will take terameprocol for 5 consecutive days each month by IV. Dose level 2= 1100mg/day. NO intrasubject dose escalation.
- Arm 3 +EIASD Level 3: subjects on the +EIASD (Level 3) treatment arm were taking one of these antiseizure drugs: phenytoin, carbamazepine, phenobarbital, primidone and oxcarbazepine.
  Subjects will take terameprocol for 5 consecutive days each month by IV. Dose level 3= 1700mg/day. NO intrasubject dose escalation. Includes pts at the new formulation TC6 at 1700mg
- Arm 4 +EIASD Level 4: subjects on the +EIASD (Level 4) treatment arm were taking one of these antiseizure drugs: phenytoin, carbamazepine, phenobarbital, primidone and oxcarbazepine.
  Subjects will take terameprocol for 5 consecutive days each month by IV. Dose level 4= 2220mg/day. NO intrasubject dose escalation.
- Arm 5 Non-Enzyme Inducing Antiseizure Drug (-EIASD) Level 1: Subjects in the -EIASD group were either not being treated with antiseizure drugs or were taking ones that did not significantly induce hepatic enzymes such as gabapentin, lamotrigine, valproic acid, levetiracetam, tiagabine, topiramate, zonisamide and felbamate.
  Subjects will take terameprocol for 5 consecutive days each month by IV. Level 1 = 750mg/day. NO intrasubject dose escalation.
  PK data will be collected on day one of cycle one infusion
- Arm 6 -EIASD Level 2: Subjects in the -EIASD group were either not being treated with antiseizure drugs or were taking ones that did not significantly induce hepatic enzymes such as gabapentin, lamotrigine, valproic acid, levetiracetam, tiagabine, topiramate, zonisamide and felbamate.
  Subjects will take terameprocol for 5 consecutive days each month by IV. Level 2 = 1100mg/day. NO intrasubject dose escalation.
  PK data will be collected on day one of cycle one infusion
- Arm 7 -EIASD Level 3: Subjects in the -EIASD group were either not being treated with antiseizure drugs or were taking ones that did not significantly induce hepatic enzymes such as gabapentin, lamotrigine, valproic acid, levetiracetam, tiagabine, topiramate, zonisamide and felbamate.
  Subjects will take terameprocol for 5 consecutive days each month by IV. Level 3 = 1700mg/day. NO intrasubject dose escalation. this Arm including pts treated at the new formulation TC6 at 1700mg
  PK data will be collected on day one of cycle one infusion
- Arm 8 -EIASD Level 4: Subjects in the -EIASD group were either not being treated with antiseizure drugs or were taking ones that did not significantly induce hepatic enzymes such as gabapentin, lamotrigine, valproic acid, levetiracetam, tiagabine, topiramate, zonisamide and felbamate.
  Subjects will take terameprocol for 5 consecutive days each month by IV. Level 4 = 2200mg/day. NO intrasubject dose escalation.
  PK data will be collected on day one of cycle one infusion
- Arm 9 - Non Stratified (Both +EIASD and -EIASD): Subjects in this group were not stratified based on anti-sezuire medication..
  Subjects will take terameprocol for 5 consecutive days each month by IV. This was for dose 2200mg/day. New formulation TC6.
Period: Overall Study
Arm/Group | Arm 1 Enzyme Inducing Antiseizure Drug (+ EIASD) Level 1 | Arm 2 +EIASD Level 2 | Arm 3 +EIASD Level 3 | Arm 4 +EIASD Level 4 | Arm 5 Non-Enzyme Inducing Antiseizure Drug (-EIASD) Level 1 | Arm 6 -EIASD Level 2 | Arm 7 -EIASD Level 3 | Arm 8 -EIASD Level 4 | Arm 9 - Non Stratified (Both +EIASD and -EIASD)
Started | 3 | 4 | 5 | 2 | 3 | 3 | 6 | 6 | 3
Completed | 3 | 3 | 5 | 2 | 3 | 3 | 6 | 6 | 3
Not Completed | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — pts declining status | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: high grade gliomas (GBM, AA or AO) histologically confirmed
Groups:
- Arm 1 +EIASD: subjects on the +EIASD treatment arm were taking one of these antiseizure drugs: phenytoin, carbamazepine, phenobarbital, primidone and oxcarbazepine.
  Subjects will take terameprocol for 5 consecutive days each month by IV. Starting dose is 750mg/day. Dose escalation is 750, 1100, 1700, 2200, 3000, 4000, 5300, 7000, and 9300. NO intrasubject dose escalation.
  PK (pharmacological study) data will be collected on day one of cycle one infusion
- Arm 2 -EIASD: Subjects in the -EIASD group were either not being treated with antiseizure drugs or were taking ones that did not significantly induce hepatic enzymes such as gabapentin, lamotrigine, valproic acid, levetiracetam, tiagabine, topiramate, zonisamide and felbamate.
  Subjects will take terameprocol for 5 consecutive days each month by IV. Starting dose is 750mg/day. Dose escalation is 750, 1100, 1700, 2200, 3000, 4000, 5300, 7000, and 9300. NO intrasubject dose escalation.
  PK (pharmacological study) data will be collected on day one of cycle one infusion
- Arm 3 no Stratification (+EIASD or -EIASD): Subjects were not stratified by antiseizure drugs
  Subjects will take terameprocol for 5 consecutive days each month by IV. Starting dose is 750mg/day. Only dose tested: 2200.
  NO intrasubject dose escalation.
  PK (pharmacological study) data will be collected on day one of cycle one infusion
- Total: Total of all reporting groups
Arm/Group | Arm 1 +EIASD | Arm 2 -EIASD | Arm 3 no Stratification (+EIASD or -EIASD) | Total
Number analyzed (Participants) | 14 | 18 | 3 | 35
Age, Continuous [Median (Full Range); unit: years] | 47 [29 to 67] | 45 [33 to 71] | 57 [36 to 65] | 46 [29 to 71]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 11 | 1 | 19
  Male | 7 | 7 | 2 | 16
Karnofsky Performance Status [Number; unit: participants] — this is a performance assessment, or functional impairment. 100% is a perfect score no impariment (highest score) and 60% Requires occasional assistance, but is able to care for most of his personal needs. You had to have at least a 60% to be eligible fof the study.
  participants
    100 | 2 | 1 | 1 | 4
    90 | 6 | 7 | 0 | 13
    80 | 0 | 5 | 0 | 5
    70 | 4 | 4 | 1 | 9
    60 | 2 | 1 | 1 | 4
Histologic diagnosis [Number; unit: participants]
  Glioblastoma | 5 | 7 | 3 | 15
  anaplastic oligodendroglioma | 5 | 5 | 0 | 10
  anaplastic astrocytoma | 4 | 6 | 0 | 10

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (Phase I)
Description: Using the PEG formulation pts both with and without enzyme inducing antiseizure drugs (EIASD) were treated at Doses 750, 1100, 1700, 2200 mg/day for five days = 28pts Using the PEG free formulation pts with and without EIASD) were treated at 1700 and 2200 mg/day X 5 days = 8pgs
Time Frame: first 30 days of treatment
Measure: Number; unit: mg/day x 5 days
Groups:
- Arm 1 +EIASD (Enzyme-inducing Antizeizure Drug): subjects on the +EIASD (Level 1) treatment arm were taking one of these antiseizure drugs: phenytoin, carbamazepine, phenobarbital, primidone and oxcarbazepine.
  Subjects will take terameprocol for 5 consecutive days each month by IV. Various Dose levels 1= 750mg/dayx5; 2=1100mg/dayx5; 3=1700mg/dayx5; 4=2200mg/dayx5
  NO intrasubject dose escalation.
  PK data will be collected on day one of cycle one infusion
- ARM 2 -EIASD (Enzyme-inducing Antizeizure Drug): Subjects in the -EIASD group were either not being treated with antiseizure drugs or were taking ones that did not significantly induce hepatic enzymes such as gabapentin, lamotrigine, valproic acid, levetiracetam, tiagabine, topiramate, zonisamide and felbamate.
  Subjects will take terameprocol for 5 consecutive days each month by IV. Various Dose levels 1= 750mg/dayx5; 2=1100mg/dayx5; 3=1700mg/dayx5; 4=2200mg/dayx5
  NO intrasubject dose escalation.
  PK data will be collected on day one of cycle one infusion
- ARM 3 (No Stratification): Subjects in this group were not stratified based on anti-sezuire medication..
  Subjects will take terameprocol for 5 consecutive days each month by IV. This was for dose 2200mg/day.
  New formulation TC6.
Arm/Group | Arm 1 +EIASD (Enzyme-inducing Antizeizure Drug) | ARM 2 -EIASD (Enzyme-inducing Antizeizure Drug) | ARM 3 (No Stratification)
Number analyzed (Participants) | 14 | 18 | 3
mg/day x 5 days | 1700 | 1700 | 1700

2. Primary Outcome: Maximum Tolerated Dose (Phase I) - Dose Limiting Toxicity (DLT)
Description: Dose limiting Toxicity defined as: Treatment related events; absolute neutrophil count </=500 /mm3; platelets count </=25,000/mm3; febrile neutropenia; any grade 3 or 4 non-hematologic toxicity; any delay in starting subsequent course of treatment for >14 days because of incomplete recovery from treatment
Time Frame: First 30 days
Population: +EIASD on hepatic enzyme-inducing drugs; -EIASE not on hepatic enzyme-induzing drug or drugs that significantly induce the hepatic enzyme.
  IV Formulations: +PEG; 10mg/mL solution of PEG 300, hydroxypropyl-B-cyclodextrin & water ; -PEG; 6mg/mL, hydroxypropyl-B-cyclodextrin & water - NEW TC6 formulation
Measure: Number; unit: Dose Limiting Toxicities (DLT)
Groups:
- + EIASD Level 1 (750 mg/dayx5D): subjects on the +EIASD (Level 1) treatment arm were taking one of these antiseizure drugs: phenytoin, carbamazepine, phenobarbital, primidone and oxcarbazepine.
  Subjects will take terameprocol for 5 consecutive days each month by IV. Dose level 1= 750mg/day. NO intrasubject dose escalation.
  PK data will be collected on day one of cycle one infusion
  +PEG Formulation
- +EIASD Level 2 (1100 mg/dayx5D): subjects on the +EIASD (Level 2) treatment arm were taking one of these antiseizure drugs: phenytoin, carbamazepine, phenobarbital, primidone and oxcarbazepine.
  Subjects will take terameprocol for 5 consecutive days each month by IV. Dose level 2= 1100mg/day. NO intrasubject dose escalation.
  PK data will be collected on day one of cycle one infusion
  +PEG Formulation
- +EIASD Level 3 (1700 mg/dayx5D): subjects on the +EIASD (Level 3) treatment arm were taking one of these antiseizure drugs: phenytoin, carbamazepine, phenobarbital, primidone and oxcarbazepine.
  Subjects will take terameprocol for 5 consecutive days each month by IV. Dose level 3= 1700mg/day. NO intrasubject dose escalation.
  PK data will be collected on day one of cycle one infusion
  +PEG Formulation; Includes patientss at the new formulation TC6 (-PEG)
- +EIASD Level 4 (2200 mg/dayx5D): subjects on the +EIASD (Level 4) treatment arm were taking one of these antiseizure drugs: phenytoin, carbamazepine, phenobarbital, primidone and oxcarbazepine.
  Subjects will take terameprocol for 5 consecutive days each month by IV. Dose level 4= 2220mg/day. NO intrasubject dose escalation.
  PK data will be collected on day one of cycle one infusion
  +PEG Formulation
- -EIASD Level 1 (750 mg/dayx5D): Subjects in the -EIASD group were either not being treated with antiseizure drugs or were taking ones that did not significantly induce hepatic enzymes such as gabapentin, lamotrigine, valproic acid, levetiracetam, tiagabine, topiramate, zonisamide and felbamate.
  Subjects will take terameprocol for 5 consecutive days each month by IV. Level 1 = 750mg/day. NO intrasubject dose escalation.
  PK data will be collected on day one of cycle one infusion
  +PEG Formulation
- -EIASD Level 2 (1100 mg/dayx5D): Subjects in the -EIASD group were either not being treated with antiseizure drugs or were taking ones that did not significantly induce hepatic enzymes such as gabapentin, lamotrigine, valproic acid, levetiracetam, tiagabine, topiramate, zonisamide and felbamate.
  Subjects will take terameprocol for 5 consecutive days each month by IV. Level 2 = 1100mg/day. NO intrasubject dose escalation.
  PK data will be collected on day one of cycle one infusion
  +PEG Formulation
- -EIASD Level 3 (1700 mg/dayx5D): Subjects in the -EIASD group were either not being treated with antiseizure drugs or were taking ones that did not significantly induce hepatic enzymes such as gabapentin, lamotrigine, valproic acid, levetiracetam, tiagabine, topiramate, zonisamide and felbamate.
  Subjects will take terameprocol for 5 consecutive days each month by IV. Level 3 = 1700mg/day. NO intrasubject dose escalation.
  PK data will be collected on day one of cycle one infusion
  +PEG Formulation and new TC6 -PEG Formulation - Pts treated from both formulations
- -EIASD Level 4 (2200 mg/dayx5D): Subjects in the -EIASD group were either not being treated with antiseizure drugs or were taking ones that did not significantly induce hepatic enzymes such as gabapentin, lamotrigine, valproic acid, levetiracetam, tiagabine, topiramate, zonisamide and felbamate.
  Subjects will take terameprocol for 5 consecutive days each month by IV. Level 4 = 2200mg/day. NO intrasubject dose escalation.
  PK data will be collected on day one of cycle one infusion
  +PEG Formulation
- Non Stratified (Both +EIASD and -EIASD): Subjects in this group were not stratified based on anti-sezuire medication..
  Subjects will take terameprocol for 5 consecutive days each month by IV. This was for dose 2200mg/day.
  New formulation TC6 - NONPEG or -PEG. (polyethylene glycol )
Arm/Group | + EIASD Level 1 (750 mg/dayx5D) | +EIASD Level 2 (1100 mg/dayx5D) | +EIASD Level 3 (1700 mg/dayx5D) | +EIASD Level 4 (2200 mg/dayx5D) | -EIASD Level 1 (750 mg/dayx5D) | -EIASD Level 2 (1100 mg/dayx5D) | -EIASD Level 3 (1700 mg/dayx5D) | -EIASD Level 4 (2200 mg/dayx5D) | Non Stratified (Both +EIASD and -EIASD)
Number analyzed (Participants) | 3 | 4 | 5 | 2 | 3 | 3 | 6 | 6 | 3
Dose Limiting Toxicities (DLT) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2

3. Secondary Outcome: Pharmacokinetics - Total Body Clearance
Description: effect of hepatic enzyme-inducing drugs on PKs
  Cycle 1 Day 1 of treatment: Predose: 1hour(hr) prior, 15minutes(min) prior; postdose: 1 hr15 min; 1.5hr, 2, 3,4, 6, 24 hrs.
  Cycle Day 5 of treatment: Predose: 1hour(hr) prior, 15minutes(min) prior; postdose: 1 hr15 min; 1.5hr, 2, 3,4, 6, 24 hrs.
Time Frame: Cycle 1 Day 1- Predose: 1hour(hr) prior, 15minutes(min) prior; postdose: 1 hr15 min; 1.5hr, 2, 3,4, 6, 24 hrs. and Cycle 1 Day 5 Predose: 1hour(hr) prior, 15minutes(min) prior; postdose: 1 hr15 min; 1.5hr, 2, 3,4, 6, 24 hrs.
Population: No PKs were collected for the three patients who were treated on Arm 3 (all EIASD). Due to incomplete collection of PKs on Cycle 1 Day 5 only the PKs from Cycle 1 Day 1 were used in the analysis
Measure: Mean (Standard Deviation); unit: Liters/hour
Groups:
- Arm 1 +EIASD: subjects on the +EIASD treatment arm were taking one of these antiseizure durgs: phenytoin, carbamazepine, phenobarbital, primidone and oxcarbazepine.
  Subjects will take terameprocol for 5 consecutive days each month by IV. Starting dose is 750mg/day. Dose escalation is 750, 1100, 1700, 2200, 3000, 4000, 5300, 7000, and 9300. NO intrasubject dose escalation.
  PK (pharmacological study) data will be collected on day one of cycle one infusion
Arm/Group | Arm 1 +EIASD | Arm 2 -EIASD
Number analyzed (Participants) | 9 | 16
Liters/hour | 53.7 (14.6) | 54.4 (20.8)
Statistical Analysis 1: Comparison: Arm 1 +EIASD vs Arm 2 -EIASD; Test type: Superiority or Other; p = 0.9, t-test, 2 sided; Mean Difference (Final Values) = 1.3

4. Secondary Outcome: Pharmacokinetics - Steady-State Apparent Volume Distribution
Description: as for outcome 3
Time Frame: as for outcome 3
Population: no PKs were collected for Arm 3. Due to incomplete collection of PKs on Cycle 1 Day 5 only the PKs from Cycle 1 Day 1 were used in the analysis
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | Arm 1 +EIASD | Arm 2 -EIASD
Number analyzed (Participants) | 9 | 16
Liters | 706 (425) | 612 (478)
Statistical Analysis 1: Comparison: Arm 1 +EIASD vs Arm 2 -EIASD; Test type: Superiority or Other; p = 0.6, t-test, 2 sided; Mean Difference (Final Values) = 15.4

5. Secondary Outcome: Pharmacokinetics - Terminal Phase Half-life
Description: effect of hepatic enzyme-inducing drugs on PKs
Time Frame: as for outcome 3
Population: no PKs for Arm 3 (All EIASD) were collected. Due to incomplete collection of PKs on Cycle 1 Day 5 only the PKs from Cycle 1 Day 1 were used in the analysis
Measure: Mean (Standard Deviation); unit: Hour
Arm/Group | Arm 1 +EIASD | Arm 2 -EIASD
Number analyzed (Participants) | 9 | 16
Hour | 18.2 (8.8) | 17.1 (9.4)
Statistical Analysis 1: Comparison: Arm 1 +EIASD vs Arm 2 -EIASD; Test type: Superiority or Other; p = 0.8, t-test, 2 sided; Mean Difference (Final Values) = 6.4

6. Secondary Outcome: Efficacy - Best Overall Response
Description: Response Criteria: Complete Response (CR): complete disappearance of all tumor, off all steroids, stable or improving neuro exam for min of 4wks; Partial Response (PR): Greater than 50% reduction in tumor size, bi-dimensional MRI/CT, stable steroids, stable or improving neuro for min of 4 wks; Progressive Disease (PD): Progressive neurologic abnormalities not explanined by causes unrelated to tumor progression, or 25% increase in size of tumor by MRI/CT scan, or if new lesion appears; Stable Disease (SD): patient whose clinical status and MRI/CT measurements do not meet the criteria for CR, PR or PD.
Time Frame: About 2 years
Population: 3 pt did not have proper scans to be evaluable for analysis
Measure: Number; unit: participants
Groups:
- Phase 1 Terameprocol: subjects were either on the +EIASD antiseizure durgs: (phenytoin, carbamazepine, phenobarbital, primidone and oxcarbazepine). or not on antiseizure drugs - or those effecting hepatic enzymes ( -EIASD) such as gabapentin, lamotrigine, valproic acid, levetiracetam, tiagavine, topiramate, zonisamide and felbamate.
  PK (pharmacological study) data will be collected on day one of cycle one infusion
Arm/Group | Phase 1 Terameprocol
Number analyzed (Participants) | 32
participants
  Complete Response | 0
  Partial Response | 0
  Progressive Disease | 23
  Stable Disease | 9

7. Secondary Outcome: Survival
Description: Survival measured from first day of treatment to date of death
Time Frame: time to death - up to 12 months
Population: 3 pts still alive at time of analysis
Measure: Median (Standard Deviation); unit: months
Arm/Group | Phase 1 Terameprocol
Number analyzed (Participants) | 32
months | 5.5 (8.4)

ADVERSE EVENTS:
Time Frame: While patients were actively on treatment and for 30 days post treatment
Groups:
- + EIASD Level 1 (750 mg/dayx5D): subjects on the +EIASD (Level 1) treatment arm were taking one of these antiseizure durgs: phenytoin, carbamazepine, phenobarbital, primidone and oxcarbazepine.
  Subjects will take terameprocol for 5 consecutive days each month by IV. Dose level 1= 750mg/day. NO intrasubject dose escalation.
  PK data will be collected on day one of cycle one infusion
  +PEG Formulation
- +EIASD Level 2 (1100 mg/dayx5D): subjects on the +EIASD (Level 2) treatment arm were taking one of these antiseizure durgs: phenytoin, carbamazepine, phenobarbital, primidone and oxcarbazepine.
  Subjects will take terameprocol for 5 consecutive days each month by IV. Dose level 2= 1100mg/day. NO intrasubject dose escalation.
  PK data will be collected on day one of cycle one infusion
  +PEG Formulation
- +EIASD Level 3 (1700 mg/dayx5D): subjects on the +EIASD (Level 3) treatment arm were taking one of these antiseizure durgs: phenytoin, carbamazepine, phenobarbital, primidone and oxcarbazepine.
  Subjects will take terameprocol for 5 consecutive days each month by IV. Dose level 3= 1700mg/day. NO intrasubject dose escalation.
  PK data will be collected on day one of cycle one infusion
  +PEG Formulation; Includes pts at the new formulation TC6 (-PEG)
- +EIASD Level 4 (2200 mg/dayx5D): subjects on the +EIASD (Level 4) treatment arm were taking one of these antiseizure durgs: phenytoin, carbamazepine, phenobarbital, primidone and oxcarbazepine.
  Subjects will take terameprocol for 5 consecutive days each month by IV. Dose level 4= 2220mg/day. NO intrasubject dose escalation.
  PK data will be collected on day one of cycle one infusion
  +PEG Formulation
- -EIASD Level 1 (750 mg/dayx5D): Subjects in the -EIASD group were either not being treated with antiseizure drugs or were taking ones that did not significantly induce hypatic enzynmes such as gabapentin, lamotrigine, valproic acid, levetiracetam, tiagavine, topiramate, zonisamide and felbamate.
  Subjects will take terameprocol for 5 consecutive days each month by IV. Level 1 = 750mg/day. NO intrasubject dose escalation.
  PK data will be collected on day one of cycle one infusion
  +PEG Formulation
- -EIASD Level 2 (1100 mg/dayx5D): Subjects in the -EIASD group were either not being treated with antiseizure drugs or were taking ones that did not significantly induce hypatic enzynmes such as gabapentin, lamotrigine, valproic acid, levetiracetam, tiagavine, topiramate, zonisamide and felbamate.
  Subjects will take terameprocol for 5 consecutive days each month by IV. Level 2 = 1100mg/day. NO intrasubject dose escalation.
  PK data will be collected on day one of cycle one infusion
  +PEG Formulation
- -EIASD Level 3 (1700 mg/dayx5D): Subjects in the -EIASD group were either not being treated with antiseizure drugs or were taking ones that did not significantly induce hypatic enzynmes such as gabapentin, lamotrigine, valproic acid, levetiracetam, tiagavine, topiramate, zonisamide and felbamate.
  Subjects will take terameprocol for 5 consecutive days each month by IV. Level 3 = 1700mg/day. NO intrasubject dose escalation.
  PK data will be collected on day one of cycle one infusion
- -EIASD Level 4 (2200 mg/dayx5D): Subjects in the -EIASD group were either not being treated with antiseizure drugs or were taking ones that did not significantly induce hypatic enzynmes such as gabapentin, lamotrigine, valproic acid, levetiracetam, tiagavine, topiramate, zonisamide and felbamate.
  Subjects will take terameprocol for 5 consecutive days each month by IV. Level 4 = 2200mg/day. NO intrasubject dose escalation.
  PK data will be collected on day one of cycle one infusion
  +PEG Formulation
- Non Stratified (Both +EIASD and -EIASD): Subjects in this group were not stratified based on anti-seizure medication..
  Subjects will take terameprocol for 5 consecutive days each month by IV. This was for dose 2200mg/day.
  New formulation TC6 - NONPEG or -PEG.
Arm/Group | + EIASD Level 1 (750 mg/dayx5D) | +EIASD Level 2 (1100 mg/dayx5D) | +EIASD Level 3 (1700 mg/dayx5D) | +EIASD Level 4 (2200 mg/dayx5D) | -EIASD Level 1 (750 mg/dayx5D) | -EIASD Level 2 (1100 mg/dayx5D) | -EIASD Level 3 (1700 mg/dayx5D) | -EIASD Level 4 (2200 mg/dayx5D) | Non Stratified (Both +EIASD and -EIASD)
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/4 | 0/5 | 0/2 | 0/3 | 0/3 | 0/6 | 2/6 | 2/3
Other Adverse Events (participants affected / at risk) | 3/3 | 4/4 | 5/5 | 1/2 | 2/3 | 3/3 | 6/6 | 3/6 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | + EIASD Level 1 (750 mg/dayx5D) (N=3) | +EIASD Level 2 (1100 mg/dayx5D) (N=4) | +EIASD Level 3 (1700 mg/dayx5D) (N=5) | +EIASD Level 4 (2200 mg/dayx5D) (N=2) | -EIASD Level 1 (750 mg/dayx5D) (N=3) | -EIASD Level 2 (1100 mg/dayx5D) (N=3) | -EIASD Level 3 (1700 mg/dayx5D) (N=6) | -EIASD Level 4 (2200 mg/dayx5D) (N=6) | Non Stratified (Both +EIASD and -EIASD) (N=3)
illeus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
interstitial nephritis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Constitutional Symptoms -other (General disorders) | 0 (0) | 0 (0) | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) — Failure to strived
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | + EIASD Level 1 (750 mg/dayx5D) (N=3) | +EIASD Level 2 (1100 mg/dayx5D) (N=4) | +EIASD Level 3 (1700 mg/dayx5D) (N=5) | +EIASD Level 4 (2200 mg/dayx5D) (N=2) | -EIASD Level 1 (750 mg/dayx5D) (N=3) | -EIASD Level 2 (1100 mg/dayx5D) (N=3) | -EIASD Level 3 (1700 mg/dayx5D) (N=6) | -EIASD Level 4 (2200 mg/dayx5D) (N=6) | Non Stratified (Both +EIASD and -EIASD) (N=3)
Seizure (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
dizziness (Nervous system disorders) | 1 (2) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 1 (1) | 0 (0)
fatigue (General disorders) | 1 (1) | 1 (5) | 1 (1) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 1 (1)
injection site reaction NOS (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
erythrodema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — localised exfoliation
nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2/2 (2) | 1 (2) | 0 (0) | 1 (1) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ataxia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
hypophosphatemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
lipase (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Right flank pain
proteinuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0)
hypertension (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
hypoalbuminemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
fecal incontinence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
urinary incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
platelet count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
rash acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 2 (3)
tremor (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
fever (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
General disorders and administration site condistions -other (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — failure to thrive
acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — interstitial nephritis
laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — pain-larynx
dehydration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
gait disturbance (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) — gait abnormal walking
anorexia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
mood alteration - euphoria (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
We were not able to complete the phase 2 portion of this study as the company had internal issues and no longer had funds to support the project. We did complete the phase I and determined the (Maxium Tolerated Dose) MTD, 1700mg/day x 5 days

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No